CLINICAL TRIAL: NCT02349022
Title: A Phase 2 Study - Comparison Of Positron Emission Tomography (PET/CT) With [89Zr]-Df-IAb2M and [111In]-Capromab Pendetide in the Detection of Prostate Cancer Pre-prostatectomy
Brief Title: Comparison of PET With [89Zr]-Df-IAb2M and [111In]-Capromab Pendetide in the Detection of Prostate Cancer Pre-Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-2M-03.00
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2016-08

CONDITIONS: Prostate Cancer
Keywords: [89Zr]Df-IAB2M; Prostate cancer; PET scan
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 89Zr-Df-IAB2M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [89Zr]Df-IAB2M (Experimental): A single intravenous infusion of 2.5 mCi of [89Zr]Df-IAB2M in a mass dose of 10 mg.
  Interventions: Radiation: [89Zr]Df-IAB2M

INTERVENTIONS:
Radiation: [89Zr]Df-IAB2M

SUMMARY:
The purpose of this study is to compare the diagnostic performance of [89Zr]-Df-IAB2M PET/CT with that of [111In]-capromab pendetide as an immuno PET tracer in the detection of prostate cancer pre-prostatectomy as confirmed by pathology.

Individuals participating in this study will have a [111In]-capromab pendetide scan, as well as a PET scan following the injection of [89Zr]-Df-IAB2M.

DETAILED DESCRIPTION:
IAB2M is an approximately 80 kDA molecular weight antibody fragment (a "Minibody") chelated with Desferroxamine and radiolabeled with 89Zr. [89Zr]-Df-IAB2M targets the extracellular domain of Prostate Membrane Specific Antigen (PSMA) expressed on most primary and metastatic prostate cancer lesions.

[111In]-capromab pendetide (Prostascint®) is an FDA approved imaging agent targeting the intracellular domain of PSMA. It is anticipated that [89Zr]-Df-IAB2M will outperform Prostascint® because of this targeting difference.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL criteria listed below for entry:

* Age ≥ 18 years
* Signed, written IRB-approved informed consent
* Patients newly diagnosed with biopsy-proven prostate cancer, thought to be a candidate for prostatectomy after standard diagnostic evaluation (e.g. chest x-ray, CT scan or MRI) who are at high-risk for pelvic lymph node metastases.
* High Risk defined as:

  * Gleason score ≥ 8 or
  * Gleason 4+3 with a PSA > 10 or
  * PSA > 20 ng/mL or
  * T3a
* Patients scheduled for a [111In]-capromab pendetide scan or had a recent [111In]-capromab pendetide scan within 28 days of screening visit or would be willing to undergo a [111In]-capromab pendetide scan
* Karnofsky Performance status of ≥ 60
* Life expectancy of at least 6 months
* Patients with any previous history of another malignancy (other than in-situ cancer, basal or squamous cell skin cancer) must be disease free for a period of three years.
* Acceptable liver function:

  * Bilirubin ≤ 1.5 times upper limit of normal or <3 x ULN for patients with Gilbert's disease
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase ≤ 2.5 times upper limit of normal (if liver metastases are present, then ≤ 5 x ULN is allowed)
* Acceptable renal function:

  * Serum creatinine within normal limits, OR
  * calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Acceptable hematologic status:

  * Granulocyte ≥ 1500 cells/mm3
  * Platelet count ≥ 150,000 (plt/mm3)
  * Hemoglobin ≥ 9 g/dL
* For men of child-producing potential, the use of effective contraceptive methods during the study

Exclusion Criteria:

Patients will be excluded from entry if ANY of the criteria listed below are met:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months
* Unstable arrhythmia, or evidence of ischemia on ECG
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy for prostate cancer.
* Unwillingness or inability to comply with procedures required in this protocol
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease (eg, hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Previous [111In]-capromab pendetide image test

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Compare sensitivity/specificity/PPV/NPV/Accuracy of [111In] capromab pendetide SPECT/CT to [89Zr]-Df-IAB2M PET/CT as confirmed by pathology | 6 weeks

SECONDARY OUTCOMES:
Assess the safety of a single dose of [89Zr]-Df-IAB2M | Day 1 through Day 13
Histopathologic correlation of PSMA expression and prostate cancer from surgical or biopsy specimens with uptake of [89Zr]-Df-IAB2M on PET/CT | Day 1 through Day 13
Compare the concordant and discordant rate for positive/negative areas of uptake between [111In]-Capromab pendetide SPECT/CT to [89Zr]-Df-IAB2M PET/CT using pathology for ground truth of disease status | Day 1 through Day 13
Compare the sensitivity/specificity/PPV/NPV/Accuracy of conventional imaging (CT/MRI/Bone scan) to [89Zr]-Df-IAB2M PET/CT using pathology for ground truth of disease status | Day 1 through Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Urology Specialists, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes